CLINICAL TRIAL: NCT05072106
Title: An Open-Label, Multicenter Study to Assess the Potential Effects of Bosentan (a Moderate CYP3A4 Inducer) on the Pharmacokinetics of Lurbinectedin (PM01183) in Patients With Advanced Solid Tumors
Brief Title: Study to Evaluate the Effect of Bosentan on the Pharmacokinetics of Lurbinectedin in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PM1183-A-019-20
Record Dates: First submitted 2021-09-02; First posted 2021-10-08 (Actual); Results first posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — PM 01183; Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single agent lurbinectedin cycle (Active Comparator): 3.2 mg/m² as a 1-hour i.v. infusion on Day 1.
  Interventions: Drug: Lurbinectedin
- Bosentan co-administration cycle (Active Comparator): * Bosentan: 125 mg (one film-coated tablet of 125 mg) orally (p.o.) twice daily in the morning and in the evening during the prior five consecutive days before the day of lurbinectedin infusion (Day 1), and once daily on Day 1 (before lurbinectedin infusion).
  * Lurbinectedin: 3.2 mg/m² as a 1-hour i.v. infusion on Day 1 in first three patients. Dose for remaining five patients will depend on PK and safety outcomes in first three patients.
  Interventions: Drug: Lurbinectedin; Drug: Bosentan

INTERVENTIONS:
Drug: Lurbinectedin — 3.2 mg/m² as a 1-hour i.v. infusion on Day 1.
  Other Names: PM01183
Drug: Bosentan — Bosentan: 125 mg (one film-coated tablet of 125 mg) orally (p.o.) twice daily in the morning and in the evening during the prior five consecutive days before the day of lurbinectedin infusion (Day 1), and once daily on Day 1 (before lurbinectedin infusion).
  Arms: Bosentan co-administration cycle

SUMMARY:
Prospective, open-label, two-way crossover, phase Ib drug-drug interaction study in patients with advanced solid tumors.

The study consisting of two lurbinectedin cycles, one cycle in combination with bosentan and one cycle as single agent (in different order depending on the study sequence), and one additional third cycle of lurbinectedin as a single agent for patients who meet the continuation criteria and obtain a clinical benefit after the first two cycles.

DETAILED DESCRIPTION:
All patients will receive a maximum of three cycles: two consecutive cycles of lurbinectedin, one cycle with and one cycle without bosentan co-administration (in different order depending on the study Sequence 1 or Sequence 2 of treatment), followed by a third cycle with lurbinectedin alone (this last optional for patients with clinical benefit). Lurbinectedin will be administered as a 1-hour intravenous (i.v.) infusion every three weeks (q3wk) via a central or peripheral vein. The dose of lurbinectedin will be 3.2 mg/m² for all patients when administered with and without bosentan. If toxicity occurs, the appropriate intra-patient dose level (DL) reductions will be implemented in the subsequent cycle.

Patients will be randomized in a 1:1 ratio to Sequence 1 (TR: Test-Reference; lurbinectedin + bosentan in Cycle 1) or Sequence 2 (RT: reference-Test; lurbinectedin + bosentan in Cycle 2).

Patients will receive lurbinectedin until disease progression, unacceptable toxicity, consent withdrawal or while it is considered to be in their best interest.

Treatment with lurbinectedin outside this study could be continued under a Compassionate Use Agreement after the completion of the optional third study cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signed and dated written informed consent prior to any specific study procedure.
2. Male or female with age ≥ 18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1.
4. Life expectancy > 3 months.
5. Pathologically confirmed diagnosis of advanced solid tumors [except for primary central nervous system (CNS) tumors], for which no approved therapy exists.
6. Recovery to grade ≤ 1 from drug-related adverse events (AEs) of previous treatments, excluding alopecia and grade ≤2 asthenia or fatigue, according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v.5).
7. Laboratory values within fourteen days prior to registration: a) Absolute neutrophil count (ANC) > 2.0 x 109/L, platelet count > 120 x 109/L and hemoglobin > 9.0 g/dL (patients may be transfused as clinically indicated prior to study entry). b) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal (ULN). c) Serum total bilirubin ≤ 1.0 x ULN. If total bilirubin is > 1.0 x ULN, but ≤ 1.5 x ULN, direct bilirubin must be ≤ 1.0 x ULN. d) Albumin ≥ 3.5 g/dL. e) Creatinine clearance (CLcr) >= 30 mL/min (using Cockcroft and Gault's formula).

   f) Creatine phosphokinase (CPK) ≤ 2.5 x ULN.
8. Left ventricular ejection fraction (LVEF) by echocardiography (ECHO) or multiple-gated acquisition (MUGA) within normal range (according to institutional standards).
9. Evidence of non-childbearing status for women of childbearing potential (WOCBP). WOCBP must agree to use a highly effective contraceptive measure up to six months after treatment discontinuation. As bosentan may render hormonal contraceptives ineffective, and taking into account the teratogenic effects observed in animals, hormonal contraceptives cannot be the sole method of contraception during treatment with bosentan. Fertile male patients with WOCBP partners should use condoms during treatment and for four months following the last investigational medicinal product (IMP) dose.

Exclusion Criteria:

1. Concomitant diseases/conditions: a) History or presence of unstable angina, myocardial infarction, congestive heart failure, or clinically significant valvular disease within last year. b) Symptomatic arrhythmia or any uncontrolled arrhythmia requiring ongoing treatment. c) Known cirrhosis, alcohol induced steatosis, or chronic active hepatitis. For hepatitis B, this includes positive test for both Hepatitis B surface antigen (HBsAg) and quantitative Hepatitis B polymerase chain reaction (PCR or HVB-DNA+). For hepatitis C, this includes positive test for both Hepatitis C antibody and quantitative Hepatitis C by PCR (or HVCRNA+). d) History of obstructive cholestatic liver disease (suitable for stenting procedure) or biliary sepsis in the past 2 months.

   e) Active COVID-19 disease (this includes positive test for SARS-CoV-2 in nasopharyngeal/oropharyngeal swabs or nasal swabs by PCR).
2. Symptomatic, progressive or corticosteroids-requiring documented brain metastases or leptomeningeal disease involvement. Patients with asymptomatic documented stable brain metastases not requiring corticosteroids during the last four weeks are allowed.
3. Use of (strong or moderate) inhibitors or inducers of CYP3A4 activity within three weeks prior to Day 1 of Cycle 1.
4. Use of CYP3A4 substrates for which concomitant administration with moderate CYP3A4 inductor is contraindicated.
5. Treatment with any investigational product within the 30 days before Day 1 of Cycle 1.
6. Women who are pregnant or breast-feeding and fertile patients (men and women) who are not using an effective method of contraception.
7. Psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pharma Mar, S.A., Study Director — PharmaMar
Locations (2):
- Spain (2):
  - Fundación Jiménez Diaz, Madrid
  - Hospital de Sanchinarro, Madrid

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11 patients were included/treated at 2 sites: 7 in Sequence 1 (TR: Test-Reference; bosentan+lurbinectedin in Cycle 1) and 4 in Sequence 2 (RT: Reference-Test; bosentan+lurbinectedin in Cycle 2). Patients participated between 14 Jan 2021 and 22 Dec 2021. The 1st dose of the 1st cycle was given on 25 Jan 2021 and the last dose of the last cycle on 25 Nov 2021
Groups:
- Sequence 1 (TR: Test-Reference): Patients received two consecutive cycles of lurbinectedin, the first one with bosentan co-administration and the second one lurbinectedin alone, followed by a third cycle with lurbinectedin alone (this last was optional for patients with clinical benefit).
- Sequence 2 (RT: Refence-Test): Patients received two consecutive cycles of lurbinectedin, the first one lurbinectedin alone and the second one with bosentan co-administration, followed by a third cycle with lurbinectedin alone (this last was optional for patients with clinical benefit)
Period: Overall Study
Arm/Group | Sequence 1 (TR: Test-Reference) | Sequence 2 (RT: Refence-Test)
Started | 7 | 4
Completed | 0 | 0
Not Completed | 7 | 4
Not completed — Progressive disease | 3 | 3
Not completed — Compassionate use | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 (TR: Test-Reference) | Sequence 2 (RT: Refence-Test) | Total
Number analyzed (Participants) | 7 | 4 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 4 | 1 | 5
Age, Continuous [Median (Full Range); unit: years] | 67 [58 to 74] | 60 [35 to 65] | 63 [35 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 3 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7 | 4 | 11
Weight [Median (Full Range); unit: kg] | 66.4 [44.3 to 83.7] | 72.4 [57.5 to 102.9] | 66.4 [44.3 to 102.9]
Height [Median (Full Range); unit: cm] | 163 [154 to 176] | 174.5 [168 to 183] | 168 [154 to 183]
Body Surface Area [Median (Full Range); unit: square metre] | 1.7 [1.5 to 2.0] | 1.9 [1.7 to 2.2] | 1.7 [1.5 to 2.2]
ECOG PS [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group Performance Status (ECOG PS) PS 0: Fully active able to carry on all pre-disease performance without restriction PS 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature PS 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours PS 3: Capable of only limited selfcare; confined to bed/chair more than 50% of waking hours PS 4: Completely disabled; cannot carry on any selfcare; totally confined to bed/chair PS 5: Dead
  Participants
    PS 0 | 4 | 2 | 6
    PS 1 | 3 | 2 | 5
Stage at diagnosis [Count of Participants; unit: Participants]
  Early | 4 | 1 | 5
  Locally advanced | 2 | 1 | 3
  Metastatic | 1 | 2 | 3
Primary tumor site [Count of Participants; unit: Participants]
  Lung | 1 | 2 | 3
  Ovarian | 1 | 1 | 2
  Breast | 1 | 0 | 1
  Cervical | 1 | 0 | 1
  Colon | 1 | 0 | 1
  Gall bladder | 1 | 0 | 1
  Mesothelioma | 1 | 0 | 1
  Neuroendocrine tumor | 0 | 1 | 1
Number of disease sites at baseline [Median (Full Range); unit: sites] | 3 [2 to 4] | 6 [2 to 7] | 3 [2 to 7]
Time from diagnosis to first infusion [Median (Full Range); unit: months] | 47.7 [30.5 to 91.6] | 13.7 [6.8 to 59.4] | 47.3 [6.8 to 91.6]
Prior surgery [Count of Participants; unit: Participants] | 7 | 2 | 9
Prior radiotherapy [Count of Participants; unit: Participants] | 4 | 4 | 8
Number of prior Anticancer Therapy lines [Median (Full Range); unit: lines] | 5 [3 to 6] | 2.5 [1 to 4] | 4 [1 to 6]
Number of prior chemotherapy lines [Median (Full Range); unit: lines] | 3 [3 to 5] | 2.5 [1 to 3] | 3 [1 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Dose-normalized Maximum Observed Plasma Concentration (Cmax) of Total Lurbinectedin: Alone and in Combination With Bosentan.
Description: Pharmacokinetic analyses will be evaluated in plasma by standard non-compartmental methods, or population methods, if necessary.
Time Frame: Preinfusion, 0.917, 1.5, 2, 3, 5, 7, 25, 49, 97 and 169 hours post lurbinectedin infusion start on Day 1 of Cycle 1 or Cycle 2 (each cycle is 21 days)
Population: Three treated patients were not evaluable for Pharmacokinetic (PK) assessments due to lack of treatment at Cycle 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/L/mg
Groups:
- Bosentan Co-administration Cycle: * Bosentan: 125 mg (one film-coated tablet of 125 mg) orally (p.o.) twice daily in the morning and in the evening during the prior five consecutive days before the day of lurbinectedin infusion (Day 1), and once daily on Day 1 (before lurbinectedin infusion).
  * Lurbinectedin: 3.2 mg/m² as a 1-hour i.v. infusion on Day 1 in first three patients. Dose for remaining five patients will depend on PK and safety outcomes in first three patients.
  Lurbinectedin: 3.2 mg/m² as a 1-hour i.v. infusion on Day 1.
  Bosentan: Bosentan: 125 mg (one film-coated tablet of 125 mg) orally (p.o.) twice daily in the morning and in the evening during the prior five consecutive days before the day of lurbinectedin infusion (Day 1), and once daily on Day 1 (before lurbinectedin infusion).
Arm/Group | Bosentan Co-administration Cycle | Single Agent Lurbinectedin Cycle
Number analyzed (Participants) | 8 | 8
μg/L/mg | 20.71 (54.81) | 21.39 (49.56)
Statistical Analysis 1: Comparison: Bosentan Co-administration Cycle vs Single Agent Lurbinectedin Cycle; Test type: Other — Bioequivalence; Least-squares geometric mean ratio = 96.83, 90% CI 2-sided [81.09 to 115.62] — The reported results are the same as the ones reported in the CSR of the trial

2. Primary Outcome: Dose-normalized Area Under the Plasma Concentration-time Profile From Time Zero to Extrapolated Infinity (AUC0-∞) of Total Lurbinectedin: Alone and in Combination With Bosentan
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Three treated patients were not evaluable for PK assessments due to lack of treatment at Cycle 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg·h/L/mg
Arm/Group | Bosentan Co-administration Cycle | Single Agent Lurbinectedin Cycle
Number analyzed (Participants) | 8 | 8
μg·h/L/mg | 58.83 (75.83) | 73.71 (86.93)
Statistical Analysis 1: Comparison: Bosentan Co-administration Cycle vs Single Agent Lurbinectedin Cycle; Test type: Other — Bioequivalence; Least-squares geometric mean ratio = 79.81, 90% CI 2-sided [64.78 to 98.32]

3. Secondary Outcome: Dose-normalized Area Under the Plasma Concentration-time Profile From Time Zero to Last Quantifiable Concentration (AUC0-t) of Total Lurbinectedin: Alone and in Combination With Bosentan
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Three treated patients were not evaluable for PK assessments due to lack of treatment at Cycle 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg·h/L/mg
Arm/Group | Bosentan Co-administration Cycle | Single Agent Lurbinectedin Cycle
Number analyzed (Participants) | 8 | 8
μg·h/L/mg | 56.33 (76.47) | 71.13 (84.97)
Statistical Analysis 1: Comparison: Bosentan Co-administration Cycle vs Single Agent Lurbinectedin Cycle; Test type: Other — Bioequivalence; Least-squares geometric mean ratio = 79.2, 90% CI 2-sided [64.12 to 97.82]

4. Secondary Outcome: Plasma Clearance (CL) of Total Lurbinectedin: Alone and in Combination With Bosentan
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Three treated patients were not evaluable for PK assessments due to lack of treatment at Cycle 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Bosentan Co-administration Cycle | Single Agent Lurbinectedin Cycle
Number analyzed (Participants) | 8 | 8
L/h | 17.00 (75.83) | 13.57 (86.93)
Statistical Analysis 1: Comparison: Bosentan Co-administration Cycle vs Single Agent Lurbinectedin Cycle; Test type: Other — Bioequivalence; Least-squares geometric mean ratio = 125.3, 90% CI 2-sided [101.71 to 154.36]

5. Secondary Outcome: Plasma Volume of Distribution at Steady-state (Vss) of Total Lurbinectedin: Alone and in Combination With Bosentan
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Three treated patients were not evaluable for PK assessments due to lack of treatment at Cycle 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Bosentan Co-administration Cycle | Single Agent Lurbinectedin Cycle
Number analyzed (Participants) | 8 | 8
L | 412.94 (78.11) | 386.69 (65.5)
Statistical Analysis 1: Comparison: Bosentan Co-administration Cycle vs Single Agent Lurbinectedin Cycle; Test type: Other — Bioequivalence; Least-squares geometric mean ratio = 106.79, 90% CI 2-sided [74.63 to 152.8]

6. Secondary Outcome: Terminal Elimination Half-life (t1/2) in Plasma of Total Lurbinectedin: Alone and in Combination With Bosentan
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Three treated patients were not evaluable for PK assessments due to lack of treatment at Cycle 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Bosentan Co-administration Cycle | Single Agent Lurbinectedin Cycle
Number analyzed (Participants) | 8 | 8
h | 35.51 (61.54) | 33.84 (35.26)
Statistical Analysis 1: Comparison: Bosentan Co-administration Cycle vs Single Agent Lurbinectedin Cycle; Test type: Other — Bioequivalence; Least-squares geometric mean ratio = 104.93, 90% CI 2-sided [69.49 to 158.44]

7. Secondary Outcome: Dose-normalized Maximum Observed Plasma Concentration (Cmax) of Unbound Lurbinectedin: Alone and in Combination With Bosentan
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Three treated patients were not evaluable for PK assessments due to lack of treatment at Cycle 2 and two patients were excluded due to extremely high unbound fraction values
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/L/mg
Arm/Group | Bosentan Co-administration Cycle | Single Agent Lurbinectedin Cycle
Number analyzed (Participants) | 6 | 6
μg/L/mg | 0.0324 (51.77) | 0.0332 (19.18)
Statistical Analysis 1: Comparison: Bosentan Co-administration Cycle vs Single Agent Lurbinectedin Cycle; Test type: Other — bioequivalence; Least-squares geometric mean ratio = 88.44, 90% CI 2-sided [65.62 to 119.19]

8. Secondary Outcome: Dose-normalized Area Under the Plasma Concentration-time Profile From Time Zero to Extrapolated Infinity (AUC0-∞) of Unbound Lurbinectedin: Alone and in Combination With Bosentan
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg·h/L/mg
Arm/Group | Bosentan Co-administration Cycle | Single Agent Lurbinectedin Cycle
Number analyzed (Participants) | 6 | 6
μg·h/L/mg | 0.095 (73.04) | 0.114 (61.09)
Statistical Analysis 1: Comparison: Bosentan Co-administration Cycle vs Single Agent Lurbinectedin Cycle; Test type: Other — bioequivalence; Least-squares geometric mean ratio = 81.8, 90% CI 2-sided [54.8 to 119.96]

9. Secondary Outcome: Dose-normalized Area Under the Plasma Concentration-time Profile From Time Zero to Last Quantifiable Concentration (AUC0-t) of Unbound Plasma Lurbinectedin: Alone and in Combination With Bosentan
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg·h/L/mg
Arm/Group | Bosentan Co-administration Cycle | Single Agent Lurbinectedin Cycle
Number analyzed (Participants) | 6 | 6
μg·h/L/mg | 0.0907 (72.73) | 0.1099 (58.24)
Statistical Analysis 1: Comparison: Bosentan Co-administration Cycle vs Single Agent Lurbinectedin Cycle; Test type: Other — bioequivalence; Least-squares geometric mean ratio = 80.26, 90% CI 2-sided [54.26 to 118.72]

10. Secondary Outcome: Plasma Clearance (CL) of Unbound Lurbinectedin: Alone and in Combination With Bosentan
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Bosentan Co-administration Cycle | Single Agent Lurbinectedin Cycle
Number analyzed (Participants) | 6 | 6
L/h | 10530.93 (73.04) | 8773.36 (61.09)
Statistical Analysis 1: Comparison: Bosentan Co-administration Cycle vs Single Agent Lurbinectedin Cycle; Test type: Other — bioequivalence; Least-squares geometric mean ratio = 123.34, 90% CI 2-sided [83.36 to 182.49]

11. Secondary Outcome: Plasma Volume of Distribution at Steady-state (Vss) of Unbound Lurbinectedin: Alone and in Combination With Bosentan
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Bosentan Co-administration Cycle | Single Agent Lurbinectedin Cycle
Number analyzed (Participants) | 6 | 6
L | 266905.87 (73.09) | 241282.16 (23.18)
Statistical Analysis 1: Comparison: Bosentan Co-administration Cycle vs Single Agent Lurbinectedin Cycle; Test type: Other — bioequivalence; Least-squares geometric mean ratio = 120.5, 90% CI 2-sided [64.79 to 224.13]

12. Secondary Outcome: Terminal Elimination Half-life (t1/2) in Plasma of Unbound Lurbinectedin: Alone and in Combination With Bosentan
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Bosentan Co-administration Cycle | Single Agent Lurbinectedin Cycle
Number analyzed (Participants) | 6 | 6
h | 37.41 (73.98) | 32.33 (39.36)
Statistical Analysis 1: Comparison: Bosentan Co-administration Cycle vs Single Agent Lurbinectedin Cycle; Test type: Other — bioequivalence; Least-squares geometric mean ratio = 120.5, 90% CI 2-sided [64.79 to 224.13]

13. Secondary Outcome: Dose-normalized Maximum Observed Plasma Concentration (Cmax) of Total Lurbinectedin Metabolite M1: Alone and in Combination With Bosentan
Description: as for outcome 1
Time Frame: Preinfusion, 0.917, 1.5, 2, 3, 5, 7 and 25 hours post lurbinectedin infusion start on Day 1 of Cycle 1 or Cycle 2 (each cycle is 21 days)
Population: Three treated patients were not evaluable for PK assessments due to lack of treatment at Cycle 2. For 1 patient all PK samples for M1 in lurbinectedin alone cycle were below the limit of quantification
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/L/mg
Arm/Group | Bosentan Co-administration Cycle | Single Agent Lurbinectedin Cycle
Number analyzed (Participants) | 8 | 7
μg/L/mg | 0.3849 (92.13) | 0.268 (78.43)
Statistical Analysis 1: Comparison: Bosentan Co-administration Cycle vs Single Agent Lurbinectedin Cycle; PK parameter used was the log-transformed metabolite/parent ratio (MPR) of M1 dose-normalized Cmax; Test type: Other — bioequivalence; Least-squares geometric mean ratio = 188.13, 90% CI 2-sided [132.93 to 266.26]

14. Secondary Outcome: Dose-normalized Area Under the Plasma Concentration-time Profile From Time Zero to Last Quantifiable Concentration (AUC0-t) of Total Lurbinectedin Metabolite M1: Alone and in Combination With Bosentan
Description: as for outcome 1
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg·h/L/mg
Arm/Group | Bosentan Co-administration Cycle | Single Agent Lurbinectedin Cycle
Number analyzed (Participants) | 8 | 7
μg·h/L/mg | 0.728 (236.22) | 0.6916 (114.55)
Statistical Analysis 1: Comparison: Bosentan Co-administration Cycle vs Single Agent Lurbinectedin Cycle; PK parameter used was the log-transformed metabolite/parent ratio (MPR) of M1 dose-normalized AUC0-t; Test type: Other — bioequivalence; Least-squares geometric mean ratio = 245.46, 90% CI 2-sided [133.4 to 451.65]

15. Secondary Outcome: Dose-normalized Maximum Observed Plasma Concentration (Cmax) of Total Lurbinectedin Metabolite M4: Alone and in Combination With Bosentan
Description: as for outcome 1
Time Frame: as for outcome 13
Population: Three treated patients were not evaluable for PK assessments due to lack of treatment at Cycle 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/L/mg
Arm/Group | Bosentan Co-administration Cycle | Single Agent Lurbinectedin Cycle
Number analyzed (Participants) | 8 | 8
μg/L/mg | 0.5617 (103.28) | 0.5528 (101.15)
Statistical Analysis 1: Comparison: Bosentan Co-administration Cycle vs Single Agent Lurbinectedin Cycle; PK parameter used was the log-transformed metabolite/parent ratio (MPR) of M4 dose-normalized Cmax; Test type: Other — bioequivalence; Least-squares geometric mean ratio = 104.94, 90% CI 2-sided [94.07 to 117.05]

16. Secondary Outcome: Dose-normalized Area Under the Plasma Concentration-time Profile From Time Zero to Last Quantifiable Concentration (AUC0-t) of Total Lurbinectedin Metabolite M4: Alone and in Combination With Bosentan
Description: as for outcome 1
Time Frame: as for outcome 13
Population: Three treated patients were not evaluable for PK assessments due to lack of treatment at Cycle 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg·h/L/mg
Arm/Group | Bosentan Co-administration Cycle | Single Agent Lurbinectedin Cycle
Number analyzed (Participants) | 8 | 8
μg·h/L/mg | 0.9962 (267.9) | 1.382 (390.96)
Statistical Analysis 1: Comparison: Bosentan Co-administration Cycle vs Single Agent Lurbinectedin Cycle; PK parameter used was the log-transformed metabolite/parent ratio (MPR) of M4 dose-normalized AUC0-t; Test type: Other — bioequivalence; Least-squares geometric mean ratio = 91.02, 90% CI 2-sided [71.39 to 116.04]

ADVERSE EVENTS:
Time Frame: From 14 January 2021 to 18 January 2022 (1 year). Adverse events will be monitored from first administration date to the end of the follow-up period which corresponds to the visit of the end of treatment (EOT), calculated as 31 days (±10 days) after the last lurbinectedin infusion or until the patient starts a new antitumor therapy or until the date of death, whichever occurs first
Arm/Group | Bosentan Co-administration Cycle | Single Agent Lurbinectedin Cycle
All-Cause Mortality (participants affected / at risk) | 1/11 | 0/8
Serious Adverse Events (participants affected / at risk) | 3/11 | 1/8
Other Adverse Events (participants affected / at risk) | 7/11 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bosentan Co-administration Cycle (N=11) | Single Agent Lurbinectedin Cycle (N=8)
Monoparesis (Nervous system disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thrombosis in device (Product Issues) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bosentan Co-administration Cycle (N=11) | Single Agent Lurbinectedin Cycle (N=8)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Monoparesis (Nervous system disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 5 (7) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review.

DOCUMENTS (2):
  • Study Protocol (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT05072106/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT05072106/SAP_001.pdf